CLINICAL TRIAL: NCT04489563
Title: Intelligent Activity-based Client-centred Training (i-ACT) in Aged Persons
Brief Title: Feasibility Study of i-ACT in Aged Persons
Acronym: i-ACT-aged
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PXL University College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: i-ACT elderly
Record Dates: First submitted 2020-07-23; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Feasibility of a Technology-based System in Aged Person
Keywords: physical activity; aged persons; technology; client-centred
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: A group of aged persons and their supervisors in day care facilities or nursing homes participated in this study to investigate the feasibility of the i-ACT system for use to engage and motivate aged persons in institutional facilities to perform physical activity. The aged persons received a 20-30 minutes test period with the self-developed programme of the i-ACT (based on hard- and software of the Microsoft Kinect). During and after the test, the feedback of the participants was noted by the supervisor (using the thinking aloud method). After the test, 3 questionnaires were conducted, i.e. the Intrinsic Motivation Inventory (IMI), System Usability Scale (SUS), and Credibility/Expectancy Questionnaire (CEQ).
  The feedback from the supervisors was also noted as part of the thinking aloud method to gather as much information as needed to adapt the prototype of the i-ACT system towards the wishes and needs from aged persons.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aged persons (Other): A feasibility test of 20-30 minutes in aged persons with an adapted Kinect-based system, i.e. i-ACT.
  Interventions: Device: i-ACT

INTERVENTIONS:
Device: i-ACT — Performing exercises with an adapted motion detection device (i.ACT) for 20-30 minutes.
  Other Names: Kinect

SUMMARY:
A mix-method cross-sectional feasibility study performed in five aged care institutes in Flanders, Belgium. A convenience sample of 48 aged persons was recruited and 12 supervisors (i.e. occupational therapy students and therapists).

Aged persons received a 20-30 minutes test with a technology-based system, i.e. intelligent Activity-based Client-centred Training system (i-ACT). The i-ACT consists of the Microsoft Kinect and adapted software in which movements can be recorded and training parameters can be set by supervisors.

During and after the test, the thinking aloud method was used. After the test, the Intrinsic Motivation Inventory, the System Usability Scale, and the Credibility/Expectancy Questionnaire were administered in the aged persons.

ELIGIBILITY:
Inclusion Criteria:

* a client of the participating centres
* cognitively able to understand and respond to questions
* follow up instructions
* understand and speak the Dutch language

Exclusion Criteria:

* severe spasticity that unables participants to perform exercises
* severe visual impairment (e.g. blindness, cataract, etc.)
* severe communication disorder that unables participants to understand and follow up instructions (e.g. aphasia, agnosia, etc.)
* persons who use electric wheelchairs who are not able to make a transfer towards a chair.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-05-12 (Actual); Study Completion 2019-05-12 (Actual)

PRIMARY OUTCOMES:
Intrinsic motivation | 30 minutes
  Using the Intrinsic Motivation Inventory to record motivational aspects
Usability of i-ACT | 10 minutes
  Using the System Usability Scale to explore the usability of i-ACT in aged persons. The System Usability Scale consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. The items scores are converted into a score from 0 (negative) to 100 (positive). A score of 72.5 or higher is considered good and above 85.0 is excellent.
Credibility/expectancy | 10 minutes
  Using the Credibility/Expectancy Questionnaire to research the credibility and expectancy of aged persons when using the i-ACT for physical activity. It is one test that consists of 2 subscales, i.e. credibility and expectancy, and scores range from 1 (totally not) to 9 (totally yes) and percentages. The percentages are converted to scores on a scale of 1 to 9/ The maximum score on each subscale is 27. A score of 13.5 is considered neutral, everything above 13.5 is positive while everything under 13.5 is considered negative.

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (5):
  - Plankeweeke, Hasselt, Limburg
  - Begralim, Riemst, Limburg
  - Begralim, Tongeren, Limburg
  - DVC H. Catharina, Zonhoven, Limburg
  - WZC H. Catharina, Zonhoven, Limburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knippenberg E, Timmermans A, Palmaers S, Spooren A. Use of a technology-based system to motivate older adults in performing physical activity: a feasibility study. BMC Geriatr. 2021 Jan 28;21(1):81. doi: 10.1186/s12877-021-02021-3. PMID 33509098